CLINICAL TRIAL: NCT01474070
Title: Influence of Discordant Intraocular Eye Pressure Readings Taken by Dynamic Contour Tonometry and Goldmann Applanation Tonometry
Brief Title: GAT-DCT-Discordance Due to Corneal Properties
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: GAT-DCT-Vergleich
Record Dates: First submitted 2011-11-03; First posted 2011-11-17 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Glaucoma
Keywords: Glaucoma; Goldmann Tonometry; Dynamic Contour Tonometry
MeSH Terms: conditions — Glaucoma | interventions — Tonometry, Ocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Intraocular Pressure Measurement — Intraocular pressure is measured with GAT and with DCT
  Other Names: Goldmann Applanation Tonometry (GAT); Dynamic Contour Tonometry (DCT)

SUMMARY:
IOP is measured with two devices (Dynamic Contour Tonometry (DCT) and Goldmann applanation tonometry (GAT)).

DETAILED DESCRIPTION:
DCT reading will be compared to a corrected GAT reading by the formula of Elsheikh, Alhasso and Pye.

* Trial with medical device

ELIGIBILITY:
Inclusion criteria:

* clinical diagnosis of glaucoma

Exclusion criteria:

* other optic neuropathy other then glaucoma
* age<18
* corneal surgery
* use of contact lenses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: glaucoma patients
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2011-11; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | IOP is measured at the only study visit
  IOP is measured with goldman-applanation tonometer and dynamic-contour-tonometer at the only study visit (V0)

SECONDARY OUTCOMES:
Demographical and clinical data | study visit V0
  Age, axial length of the eye, central corneal thickness

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kniestedt, MD, Principal Investigator — University Hospital Zurich, Ophthalmic Clinic
Locations (1):
- University Hospital Zurich, Ophthalmic Clinic, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wachtl J, Toteberg-Harms M, Frimmel S, Roos M, Kniestedt C. Correlation Between Dynamic Contour Tonometry, Uncorrected and Corrected Goldmann Applanation Tonometry, and Stage of Glaucoma. JAMA Ophthalmol. 2017 Jun 1;135(6):601-608. doi: 10.1001/jamaophthalmol.2017.1012. PMID 28494071